CLINICAL TRIAL: NCT05367713
Title: Bone Flap Osteomyelitis Following Craniectomy : Retrospective Evaluation of Clinical Presentation, Microbiological Diagnosis and Management
Acronym: BoFOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 682
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Osteitis; Cranial Flap
Keywords: Osteitis; cranial flap
MeSH Terms: conditions — Osteitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having had an osteitis of the cranial flap after craniectomy
  Interventions: Other: patients having had an osteitis of the cranial flap after craniectomy

INTERVENTIONS:
Other: patients having had an osteitis of the cranial flap after craniectomy — description of management and failure of cranial flap after craniectomy

SUMMARY:
Osteitis of the cranial flap after craniectomy is an unknown complex osteoarticular infection and there are few data concerning its epidemiology, its risk factors, and its management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cranial flap osteitis after craniectomy
* Patients who did not object to participating in the study
* Adult patients

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cranial flap osteitis after craniectomy, treated at CRIOAc Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
rate of cranial flap osteitis after craniectomy | between 2010 and 2021
  proportion of patients

SECONDARY OUTCOMES:
rate of failure in management of cranial flap osteitis after craniectomy | between 2010 and 2021
  proportion of patients having a failure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: website of CRIOAc Lyon — https://www.crioac-lyon.fr/en/